CLINICAL TRIAL: NCT01566136
Title: An Inpatient Rehabilitation Model of Care Targeting Patients With Cognitive
Brief Title: An Inpatient Rehabilitation Model of Care Targeting Patients With Cognitive Impairment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CIHR DPA-93049
Record Dates: First submitted 2012-03-21; First posted 2012-03-29 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Hip Fracture
Keywords: hip fracture patients; cognitive impairment; rehabilitation model of care
MeSH Terms: conditions — Hip Fractures; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Current routine rehab care for persons with a hip fracture and CI lacks a well integrated care system within the local hospital network. The usual approach to care at the two sites differ in one major way: patients presenting with a hip fracture to Site 1 receive surgery locally, while those presenting to Site 2 receive surgery at a different hospital because of the absence of an operating suite at this site. Within 2 to 10 days 95% of patients presenting to either site hospital's emergency room with a hip fracture, receive internal fixation or arthroplasty surgery. Patients, including some with mild and moderate CI, are then transferred to in-patient rehabilitation beds at Site 1 or Site 2. Screening of patients for dementia or delirium is not routinely done.
- Rehabilitation Model of Care (Experimental): Staff will be introduced to five components of the Patient-Centred Rehabilitation Model of Care (PCRM-CI) in a one-day workshop prior to implementing the PCRM-CI model. They will then be provided with eight additional educational sessions throughout the year. A manual detailing all aspects of training, including specifics on how to present the material, ideas for stimulating discussion, and case vignettes to illustrate training concepts was developed for our pilot study and will be used here. We also produced a short video on care of elderly with CI in rehabilitation which will be utilized in the training session. The model will be tested over a one year period with a sustainability plan in place developed by the local hospital network and the two study sites.
  Interventions: Behavioral: Rehabilitation Model of Care

INTERVENTIONS:
Behavioral: Rehabilitation Model of Care — The PCRM-CI model includes the following 5 components: rehabilitation management; dementia management; delirium prevention and management; staff education and support; and family/significant other support and education.
  Other Names: Patient Centred Rehabilitation Model of Care
  Arms: Rehabilitation Model of Care

SUMMARY:
Hip fractures are a danger to an individual's mobility, independence and ability to live in the community. When patients have a cognitive impairment (such as dementia or delirium) they do not recover as well or go back to their homes as often as those patients who do not have a cognitive impairment. Therefore, our team developed a rehabilitation model to care for patients with hip fractures, and specifically for those patients with CI. The model of care is called the Patient Centred Rehabilitation Model of Care (PCRM-CI). This 3 year study will focus on comparing the new model with usual rehabilitation care. This study will also focus on understanding the factors that could influence the use of the model on new rehabilitation units. The investigators hypothesize that patients who have received the new model of care will have better mobility outcomes over time. The investigators will collect data in 2 hospitals, 70 patients receiving the usual care and 70 patients receiving the care in the new model. The team will invite 60 staff and their unit managers as well. This study will help decision makers to use research findings to make better decisions about care of older Canadians.

DETAILED DESCRIPTION:
Background: A hip fracture is often a catastrophic event that is a significant threat to an individual's mobility, independence and ability to live in the community. Projections indicate that the incidence of hip fracture will increase nearly four-fold by 2041 in Canada. The course and outcomes of hip fracture patients are often complicated by the presence of dementia and delirium, referred to as cognitive impairment (CI), which limits access to in-patient rehabilitation. In response to this concern, members of our team developed an in-patient rehabilitation model of care for patients with hip fractures, with specific components of the model targeting patients with CI (PCRM-CI). The pre-clinical and phase I testing of the model has been completed, and preliminary evidence exists that patients with and without CI can regain their mobility and function and return to previous living arrangement at discharge from rehabilitation. This proposed 3 year study focuses on phase II, that is, to compare the PCRM-CI with usual rehabilitation care and to gain a better understanding of factors influencing implementation of the model. Decision-making partners for this proposal have identified service gaps within their local health region related to rehabilitation care of patients with hip fractures and are committed to sustaining the model beyond this study. This proposed research addresses the mandate of the current funding opportunity by improving the mobility of cognitively impaired elders, and by enhancing the capacity of research users to apply research evidence in decisions on models of care that can contribute to improved mobility for aging older Canadians.

Research Objectives: Primary Objective: To determine whether, compared to usual care, an inpatient rehabilitation model of care targeting community dwelling individuals with hip fracture and CI (dementia and/or delirium) results in improved mobility at the time of discharge from inpatient rehabilitation.

Secondary Objectives: 1) To determine if the use of the PCRM-CI for persons with hip fracture and CI will result in: i) improved mobility at 6 months post-surgery; ii) greater improvement in physical functioning at the time of discharge from inpatient rehabilitation and at 6 months post-surgery; iii) a higher proportion of patients with hip fracture returning to their previous living situation in the community at discharge and at 6 months post-surgery. 2) To determine whether the PCRM-CI results in similar improvements in mobility at discharge and 6 months post-surgery for patients with and without CI. 3) To evaluate whether the PCRM-CI improves health care providers' (HCPs) attitudes, knowledge, satisfaction and stress. 4) To examine the processes by which the PCRM-CI is implemented.

Design: A non-equivalent pre-post design will be used to evaluate the PCRM-CI as compared to usual care. All community dwelling (retirement or home) patients following a hip fracture will be eligible to participate. Two facilities will be involved in the study as multi site sampling increases robustness by allowing for comparison and contrast between sites. Study accrual will take about 16 months to complete recruitment and data collection of 70 hip fracture patients in the usual care cohort and 70 patients in the PCRM-CI cohort, based on sample size and attrition estimation from phase I. The investigators will recruit 60 HCPs and their unit managers in the study.

Methods: Baseline data will be collected within 3 days of admission to rehabilitation. Follow-up occurs within 3 days of discharge from rehabilitation and 6 months post-surgery. Patient evaluations will include mobility (mobility and locomotion items of FIMM), physical function (motor-FIM), and living arrangement (collaterals' informants reply). Other variables influencing outcomes that will be collected from the patient include: sex, co-morbidities, age, patients' level of education, social support (live alone, with spouse, or with other), pre fracture status (OARS), and pre-cognitive status (IQCODE). During the patients' stay in rehabilitation, data on dementia (MMSE), delirium screening (CAM) and severity (Delirium Index) will be collected. Lastly, focus groups with HCPs and semi-structured interviews with unit managers will be conducted, and the investigators will collect additional data through intervention logs, and field notes to examine factors influencing the model implementation.

Significance: With the aging of the population, this research will contribute to meeting the emerging health needs of Canadians by improving the provision of services for elders with CI.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older,
* admitted to rehabilitation directly from an acute care hospital after receiving surgery for a hip fracture
* living in the community, home or residential setting (where an individual has services and supports but does not require 24 hour nursing care) prior to sustaining the hip fracture,
* able to speak and understand English
* have a family member or close friend who is familiar with the patients' pre-fracture condition and can act as a collateral informant.

Exclusion Criteria:

* they have a pathologic hip fracture
* the hip fracture is associated with multiple trauma
* they have had a previous hip fracture.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mobility at 6 months | Baseline to 6 months post-surgery

SECONDARY OUTCOMES:
Change from baseline in physical functioning at 6 months | Baseline to 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Katherine S McGilton, PhD, Principal Investigator — UHN-Toronto Rehab
Locations (1):
- Northumberland Hospital, Cobourg, Ontario, Canada

REFERENCES:
- [Derived] McGilton KS, Davis AM, Naglie G, Mahomed N, Flannery J, Jaglal S, Cott C, Stewart S. Evaluation of patient-centered rehabilitation model targeting older persons with a hip fracture, including those with cognitive impairment. BMC Geriatr. 2013 Dec 13;13:136. doi: 10.1186/1471-2318-13-136. PMID 24330470
- [Derived] McGilton KS, Davis A, Mahomed N, Flannery J, Jaglal S, Cott C, Naglie G, Rochon E. An inpatient rehabilitation model of care targeting patients with cognitive impairment. BMC Geriatr. 2012 May 25;12:21. doi: 10.1186/1471-2318-12-21. PMID 22631877